CLINICAL TRIAL: NCT03403101
Title: A Phase II, Single Arm, Open Label Study to Evaluate the Efficacy and Safety of the Combination of S-1, Irinotecan and Oxaliplatin (SIRIOX) in Treating Patients With Advanced Inoperable or Metastatic Pancreatic Cancer
Brief Title: The Combination Chemotherapy of SIRIOX as First- or Second-Line Chemotherapy for Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Director, Head of Otolaryngology, Principal Investigator, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-020
Record Dates: First submitted 2017-11-28; First posted 2018-01-18 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — S 1 (combination); Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIRIOX regimen (Experimental): 5-FU and leucovorin in the FOLFIRINOX regimen were replaced with oral S-1, forming the SIRIOX regimen(S1 plus irinotecan and oxaliplatin)
  Interventions: Drug: S1; Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: S1 — Patients are planned to receive the SIRIOX regimen including S-1 (BSA < 1.2m2, 40 mg/day; BSA = 1.2~1.4 m2, 60 mg/day; BSA = 1.4~1.6 m2, 80 mg/day; BSA > 1.6 m2, 100 mg/day; oral twice daily on days 1-7, days 15-21）of every cycle.
  • 28 days a cycle.
Drug: Oxaliplatin — Patients are planned to receive the SIRIOX regimen including Oxaliplatin (OXA, 85 mg/m2; d1,d15) of every cycle.
  • 28 days a cycle
Drug: Irinotecan — Patients are planned to receive the SIRIOX regimen including Irinotecan (IRI, 180mg/m2; day 1,day 15) of every cycle.
  • 28 days a cycle

SUMMARY:
Pancreatic cancer represents the most lethal of the common malignancies with a 5-year survival rate of less than 5%. For patients who are eligible for potentially curative resection, despite mortality and morbidity rates after surgery have improved, the recurrence rate is up to 85% within 2 years. FOLFIRINOX (fluoropyrimidine/leucovorin plus irinotecan and oxaliplatin) has been proved to significantly improve the prognosis and is recommended as first line treatment in patients with advanced pancreatic cancer. However, the regimen is limited due to the severe adverse effects. Thus, the investigators replaced 5-FU and leucovorin in the FOLFIRINOX regimen with oral S-1, a new oral ﬂuoropyrimidine derivative which was proved to be the well-tolerated and effectively in large III phase randomized clinical trial, to form the SIRIOX regimen. A phase I clinical trial from Japan found that SOXIRI (S-1, oxaliplatin and irinotecan) works in patients with advanced pancreatic cancer. In this study, the researchers intend to investigate the activity and safety of the combination of this regimen in patients with advanced pancreatic cancer, as first- or second-line chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer (mainly pancreatic ductal adenocarcinoma, PDAC) is a disease with extremely poor prognosis, and is often fatal. Surgical resection is the only potentially curative technique for management of PDAC, but only approximately 15% to 20% of patients are candidates for pancreatectomy at the time of diagnosis Gemcitabine (Gem) is widely used as a standard chemotherapeutic agent for advanced pancreatic cancer. FOLFIRINOX (fluoropyrimidine/leucovorin plus irinotecan and oxaliplatin), compared with Gem, has been proved to significantly improve the objective response rate (31.6% VS. 9.4%, P < 0.001) and prolong the median survival time (11.1 months VS. 6.8 months, P < 0.001) for patients with metastatic pancreatic ductal adenocarcinoma(PDAC), who had a performance status of ECOG 0-1 score. However, it is undeniable that the adverse effects of FOLFIRINOX are severe. For example, the incidence of 3/4 grade neutrophil decrease in patients receiving FOLFIRINOX is significantly higher than those with Gem (45.7% VS. 21%, P < 0.001). Thus, it is difficult for many patients to receive standard FOLFIRINOX and benefit from the protocol. Therefore, the investigators aim to explore an improvement program of FOLFIRINOX, hoping to better benefit patients.

S-1 is a new oral fluoropyrimidine derivative in which tegafur is combined with two 5-chloro-2, 4-dihydroxypyridine modulators and oteracil potassium, a potentiator of 5-ﬂuorouracil's (5-FU's) antitumor activity that also decreases gastrointestinal toxicity. Combination chemotherapy with Gem and S-1 is reportedly well tolerated and benefits patients with advanced PDAC. Based on the results of the GEST study, S-1 is found to be non-inferior to Gem in patients' survival.

Therefore, in this study, the investigators replaced 5-FU and leucovorin in the FOLFIRINOX regimen with oral S-1, forming a SIRIOX regimen to treat patients with advanced pancreatic cancer, as first- or second-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 - 75 years old at the time of signing the ICF.
2. Patients with pathologically proved adenocarcinoma of pancreatic cancer and diagnosed with inoperable/metastatic disease (previous systemic chemotherapy, neoadjuvant or adjuvant are acceptable without Irinotecan, Oxaliplatin, or S1).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Adequate hematologic function defined as: absolute neutrophil count (ANC) >= 2,000/μL; platelets count >= 100,000/μL; hemoglobin must be >= 10 g/dL (can be corrected by growth factor or transfusion).
5. Adequate hepatic function defined as: serum bilirubin =< 1.5-fold upper limit of normal (ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) =< 3-fold ULN (5-fold ULN if liver metastasis is observed).
6. Adequate renal function with: serum creatinine =< 1.3 mg/dL or calculated creatinine clearance >= 60 mL/minute according to the Cockcroft and Gault formula.
7. At least one measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
8. Life expectancy over 12 weeks.
9. Women must be either of non-child bearing potential, or women with child-bearing potential agree to use effective a highly contraceptive method or a contraceptive implant, exception of hormonal contraception (estrogen/progesterone), during treatment from time of Screening Visit and after cessation of therapy at least 3 months.
10. Willing and able to comply with all aspects of the treatment protocol.
11. Provide written informed consent.

Exclusion Criteria:

1. Patients who are unwilling or unable to comply with the study protocol;
2. Existing anticancer treatment-related toxicities of Grades >= 2 (except for alopecia and neuropathy) according to Common Terminology Criteria for Adverse Events (CTCAE v4.03).
3. Simultaneously using targeted therapies, such as Erlotinib, Nimotuzumab etc;
4. Any severe or uncontrolled systemic disease (e.g., unstable or decompensated breathing, heart, liver or kidney disease, HIV infection, hypertension, severe arrhythmia, diabetes mellitus, massive active bleeding);
5. Large operations were performed within 14 days before entering the study, or there were surgical incisions that were not completely healed;
6. Women who are pregnant or breastfeeding;
7. Ascertained hypersensitivity to investigational product, Oxaliplatin, Irinotecan, and S1 or any of the excipients used in the study.
8. History of other malignancies within 5 years, except for adequately treated basal cell carcinoma or squamous cell carcinoma or carcinoma in situ;
9. Obvious gastrointestinal injury history, the researchers estimate may significantly affect the absorption of S1 on the whole, including the ability to swallow drugs;
10. Other combinations of anticancer therapies (including LHRH agonists, anticancer herbs, immunotherapy), except steroid hormones;
11. Patients with UGT1A1 mutations or congenital disease lack of UGT1A1 expression (e.g. Crigler-Najjar syndrome and Gilbert syndrome);
12. Patients with DPD enzyme deficiency.
13. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation, psychiatric disorder, with any other serious diseases/medical history.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 6 weeks (1.5 cycle)
  The time from the beginning of randomization to the earliest date of confirmation of tumor progression or the patient death for any reason. If the above criteria are not reached, the date of the last evaluation will be used.

SECONDARY OUTCOMES:
objective response rate (ORR) | 6 weeks (1.5 cycle)
  The proportion of patients whose tumors shrink to a certain amount for a certain period of time and include cases of complete response (CR) and partial response (PR). Calculated as: (CR cases + PR cases) / FAS × 100 (%); FAS (full analysis set) refers to the case of qualified patients, administered more than one case.
  Tumor remission rates are calculated according to the RECIST guidelines (version 1.1)
overall survival (OS) | through study completion, an average of 18 months
  The time from the beginning of randomization to the earliest date of confirmation of the patient death for any reason.
Toxicity evaluated according to the Common Terminology Criteria Adverse Events | every week
  Toxicity is evaluated according to the Common Terminology Criteria Adverse Events Version3.0,CTCAEv3.0

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, M.D., Ph.D., Study Chair — 270 Dong An Road, Shanghai 200032, China
Locations (2):
- China (2):
  - Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality
  - Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University; 270 Dong An Road, Shanghai 200032, China, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided